CLINICAL TRIAL: NCT00644449
Title: A Multicenter, Randomized, Double-Blind, Double-Dummy Comparative Trial of Azithromycin SR Versus Levofloxacin for the Treatment of Acute Exacerbation of Chronic Bronchitis (AECB)
Brief Title: A Multicenter, Randomized, Double-Blind, Double-Dummy Trial of Azithromycin SR Compared With Levofloxacin for the Treatment of Acute Symptoms of Chronic Bronchitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0661102
Record Dates: First submitted 2008-03-19; First posted 2008-03-26 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: Bronchitis, Chronic
MeSH Terms: conditions — Bronchitis, Chronic | interventions — Azithromycin; Levofloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Other: placebo; Drug: azithromycin SR (Zithromax; compound: CP-62,993)
- 2 (Experimental)
  Interventions: Other: placebo; Drug: levofloxacin

INTERVENTIONS:
Other: placebo — placebo
  Arms: 1
Drug: azithromycin SR (Zithromax; compound: CP-62,993) — azithromycin 2.0 g by mouth in the form of a slurry for 1 dose
  Arms: 1
Other: placebo — placebo
  Arms: 2
Drug: levofloxacin — 500 mg (two 250 mg capsules) by mouth once daily for 7 days
  Arms: 2

SUMMARY:
This study was performed to confirm that a single 2.0-g dose of azithromycin SR is at least as effective as 7 days of levofloxacin 500 mg/day in adults with acute exacerbation of chronic bronchitis Secondary objectives: To assess safety and the bacteriologic efficacy of both treatment regimens

ELIGIBILITY:
Inclusion Criteria:

Adult patients with a history of chronic bronchitis (i.e., chronic cough and sputum production on most days for 3 consecutive months for more than 2 years) and current evidence of an acute bacterial exacerbation of their disease, as demonstrated by production of purulent sputum and the presence of at lest 2 of the following signs and symptoms, were included: increased sputum production, increased dypsnea, increased cough, or increased sputum purulence.

Exclusion Criteria:

Key exclusion criteria were treatment with any systemic antibiotic within the previous 7 days, or the likelihood of receiving other systemic antibiotics during participation in the study; a chest radiograph consistent with pneumonia; and previously diagnosed conditions which tend to mimic or complicate the course and evaluation of the infectious process (e.g., bronchiectasis, lung abscess or empyema, active TB, pulmonary malignancy, cystic fibrosis).

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 551 (Actual)
Dates: Start 2003-01; Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
sponsor assessment of clinical response in the Clinical Per Protocol population | Test of Cure (TOC) visit (Day 14-21)

SECONDARY OUTCOMES:
investigator assessment of clinical response in the Clinical Per Protocol population | TOC visit
bacteriological response on a per pathogen basis for the Bacteriological Per Protocol population | TOC visit
sponsor assessment of clinical response in the Clinical Per Protocol population | Long-Term Follow-Up (LTFU) visit (Day 28-35)
Summary of baseline susceptibilities | Study Endpoint
adverse events | Continuous
clinical laboratory tests | Baseline and EOT visit
sponsor assessment of clinical response in the Clinical Per Protocol population | End of Treatment (EOT) visit (Day 8-11)
sponsor assessment of clinical response in the remaining study populations | TOC visit
sponsor assessment of clinical response by baseline pathogen for the Bacteriological Per Protocol population | EOT visit and TOC visit

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (61):
- United States (24):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Columbiana, Alabama
  - Pfizer Investigational Site, Tallassee, Alabama
  - Pfizer Investigational Site, Mesa, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Tempe, Arizona
  - Pfizer Investigational Site, Daytona Beach, Florida
  - Pfizer Investigational Site, Merritt Island, Florida
  - Pfizer Investigational Site, Austell, Georgia
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Madisonville, Kentucky
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Royal Oak, Michigan
  - Pfizer Investigational Site, Olive Branch, Mississippi
  - Pfizer Investigational Site, Elkhorn, Nebraska
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Allentown, Pennsylvania
  - Pfizer Investigational Site, Harrisburg, Pennsylvania
  - Pfizer Investigational Site, Morrisville, Pennsylvania
  - Pfizer Investigational Site, Willow Grove, Pennsylvania
  - Pfizer Investigational Site, Milan, Tennessee
  - Pfizer Investigational Site, San Antonio, Texas
- Brazil (3):
  - Pfizer Investigational Site, Curitiba, Paraná
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, Santo André, São Paulo
- Canada (7):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Sydney, Nova Scotia
  - Pfizer Investigational Site, Hawkesbury, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Ste-Foy, Quebec
  - Pfizer Investigational Site, North Battleford, Saskatchewan
  - Pfizer Investigational Site, Saskatoon, Saskatchewan
- Costa Rica (6):
  - Pfizer Investigational Site, Desamparados, Provincia de San José
  - Pfizer Investigational Site, Guadalupe, Provincia de San José
  - Pfizer Investigational Site, Pavas, Provincia de San José
  - Pfizer Investigational Site, Pinares de Curridabat, Provincia de San José
  - Pfizer Investigational Site, San José, Provincia de San José
  - Pfizer Investigational Site, Uruca, Provincia de San José
- Germany (2):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Rathenow
- India (6):
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Elamakkara, Cochin, Kerala
  - Pfizer Investigational Site, Indore, Madhya Pradesh
  - Pfizer Investigational Site, Pune, Maharashtra
  - Pfizer Investigational Site, Ludhiana, Punjab
  - Pfizer Investigational Site, Coimbatore, Tamil Nadu
- Lithuania (3):
  - Pfizer Investigational Site, Alytus
  - Pfizer Investigational Site, Klaipėda
  - Pfizer Investigational Site, Vilnius
- Pfizer Investigational Site, Monterrey, Nuevo León, Mexico
- Pfizer Investigational Site, Eindhoven, Netherlands
- Russia (2):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Smolensk
- Spain (2):
  - Pfizer Investigational Site, Madrid
  - Pfizer Investigational Site, Málaga
- United Kingdom (3):
  - Pfizer Investigational Site, Atherstone, Warwickshire
  - Pfizer Investigational Site, Leeds, West Yorkshire
  - Pfizer Investigational Site, Glasgow
- Pfizer Investigational Site, Caracas, Venezuela

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661102&StudyName=A%20Multicenter%2C%20Randomized%2C%20Double-Blind%2C%20Double-Dummy%20Trial%20of%20Azithromycin%20SR%20Compared%20with%20Levofloxacin%20for%20the%20Treatment%20of%20Acute%20S